CLINICAL TRIAL: NCT01453946
Title: A Multicenter, Open Label, Non-comparative Study to Evaluate the Safety of Entocort EC as a Maintenance Treatment for Crohn's Disease in Paediatric Subjects Aged 5 to 17 Years, Inclusive
Brief Title: Safety and Maintenance Study of Entocort for Children With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9422C00002
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide

ARMS (1):
- Entocort (Other): Study Medication
  Interventions: Drug: Entocort

INTERVENTIONS:
Drug: Entocort — Entocort capsules, taken orally, 6 mg daily.

SUMMARY:
A Safety for Maintenance of Entocort EC for children with mild to moderate Crohn's Disease.

DETAILED DESCRIPTION:
A Multicenter, Open label, Non-comparative Study to Evaluate the Safety of Entocort EC as a Maintenance Treatment for Crohn's Disease in Paediatric Subjects Aged 5 to 17 Years, Inclusive

ELIGIBILITY:
Inclusion Criteria:

* All male and female subjects must be aged 5 to 17, inclusive, and must not have reached their 18th birthday by the estimated final office visit.
* All subjects must weight >= 15 kg at the time of enrollment.
* Subjects must have been diagnosed and treated for active Crohn's disease of the ileum and/or ascending colon confirmed by endoscopic and/or radiographic evidence, and/or evidence of mucosal erosions and/or histology and have a PCDAI <= 10

Exclusion Criteria:

* Subjects who have had any previous intestinal resection proximal to and including the ascending colon.
* Subjects with evidence of active Crohn's disease (PCDAI > 10) and/or stricturing, prestenotic dilatation, clinical evidence of obstruction, perirectal abscess, perirectal disease with active draining fistulas, perforation, or any septic complications.
* Subjects with morning cortisol level <150 nmol/l (5.4 ug/dl) or DHEA-S below normal range for age and gender (NOTE: Subjects from the induction protocol with abnormal morning cortisol/DHEA-S levels at Visit 4, who otherwise meet the eligibility criteria, may be enrolled if the investigator decides that Entocort 6 mg is an appropriate therapy option.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohen, MD, Principal Investigator — Children's Center for Digestive Healthcare, LLC, Atlanta, Georgia, USA; Stefan Eklund, MD, Study Director — AstraZeneca Pharmaceuticals, Mölndal, Sweden
Locations (19):
- United States (7):
  - Research Site, Atlanta, Georgia
  - Research Site, Oak Lawn, Illinois
  - Research Site, Newton, Massachusetts
  - Research Site, Saint Paul, Minnesota
  - Research Site, Mays Landing, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Houston, Texas
- Canada (2):
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
- Germany (2):
  - Research Site, München
  - Research Site, Nuremberg
- Italy (3):
  - Research Site, Florence
  - Research Site, Messina
  - Research Site, Roma
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- [Derived] Cohen SA, Aloi M, Arumugam R, Baker R, Bax K, Kierkus J, Koletzko S, Lionetti P, Persson T, Eklund S. Enteric-coated budesonide for the induction and maintenance of remission of Crohn's disease in children. Curr Med Res Opin. 2017 Jul;33(7):1261-1268. doi: 10.1080/03007995.2017.1313213. Epub 2017 Apr 19. PMID 28420280
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=649&filename=ADMIRe_D9422C00002_CTD_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, 55 patients were enrolled but only 50 fulfilled the enrolment criteria.
Pre-assignment Details: 55 patients were enrolled but only 50 received treatment.
Groups:
- Entocort: Entocort 6 mg/day
Period: Overall Study
Arm/Group | Entocort
Started | 50
Completed | 41
Not Completed | 9
Not completed — Did not receive drug for the taper phase | 1
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Entocort
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 13.8 [8 to 17]
Age, Customized [Number; unit: participants]
  <=8 years | 2
  >8 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45
  Black or african american | 2
  Other | 3

OUTCOME MEASURES:

1. Secondary Outcome: PCDAI
Description: Pediatric Crohn's Disease Activity Index. The scale ranges from 0 (no activity) to 100 (high activity)
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Entocort
Number analyzed (Participants) | 49
Scores on a scale
  Baseline | 4.9 (3.6)
  Change after 12 weeks | 2.0 (7.0)
  12 weeks | 6.9 (8.1)

2. Secondary Outcome: IMPACT 3
Description: IMPACT-III - A QUALITY OF LIFE QUESTIONNAIRE FOR CHILDREN WITH INFLAMMATORY BOWEL DISEASE
Time Frame: 12 weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | Entocort
Number analyzed (Participants) | 50
Score units
  Baseline | 146.6 (12.4)
  Change after 12 weeks | 1.2 (8.6)
  12 weeks | 147.0 (15.5)

3. Primary Outcome: Adverse Event
Description: Any kind of adverse event
Time Frame: 16 weeks
Population: Safety analysis set
Measure: Number; unit: Subjects
Arm/Group | Entocort
Number analyzed (Participants) | 50
Subjects | 37

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: 12 weeks on 6 mg/day followed by 2 weeks on 3 mg/day and 2 weeks without active drug
Arm/Group | Entocort
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 36/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entocort (N=50)
Crohn's disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal haemhorrage (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entocort (N=50)
Abdominal pain (Gastrointestinal disorders) | 8
Crohn's disease (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Haematochizia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Acne (Skin and subcutaneous tissue disorders) | 6
Hirsutism (Skin and subcutaneous tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 3
Irritability (General disorders) | 4
Mood swings (Psychiatric disorders) | 4
Headache (Nervous system disorders) | 2
Cushingoid (Endocrine disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No